CLINICAL TRIAL: NCT02145208
Title: One-arm, Multi-center, International Prospective Study to Assess the Efficacy of Medi-Tate Temporary Implantable Nitinol Device (iTindTM) in Subjects With Benign Prostatic Hypertrophy (BPH).
Brief Title: Study to Assess the Efficacy of Medi-Tate iTind Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medi-Tate Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-02
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
Keywords: BPH
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: iTind
Oversight: Data Monitoring Committee: No

ARMS (1):
- Medi-Tate iTind (Experimental): TIND System
  Interventions: Device: TIND System

INTERVENTIONS:
Device: TIND System — An implant

SUMMARY:
The study will include an implantation of the iTind device and 4 follow up visits up to 12 months after the implantation.

DETAILED DESCRIPTION:
After screening , eligible patients will undergo an an implantation procedure (operative), using the iTind device.

Implantation will be performed according to the Instructions For Use.

Between the 5th - 7th days, the iTind will be retrieved through a rigid cystoscope sheath, under direct vision. Before retrieval the subject will be asked for subjective discomfort evaluation and level of urgency in the past days after device insertion, about any AE and then the device will be retrieved.

The next visits will be at 4 weeks (post device retrieval), 3 months, 6 months, and 12 months post implantation with an optional extension of follow up period (up to 36 months). In the visits the following will be assessed: Uroflow and residual urine volume tests, AE recording, IPSS, and Questions on sex performing capability and ejaculation filled out by the subjects, in the local languages.

ELIGIBILITY:
Inclusion Criteria:

* Subject signed informed consent prior to the performance of any study procedures.
* Male with symptomatic BPH. IPSS symptom severity score above 10. Peak urinary flow of below 12 ml/sec
* Prostate volume below 75 ml
* Blood CBC and biochemistry up to two weeks before screening demonstrating: Normal values of the PT, PTT and INR tests (anticoagulants should be stopped according to GCP)
* Subject that able to complete the study protocol.
* Normal Urinalysis and urine culture

Exclusion Criteria:

* cardiac arrhythmias, cardiac disease including congestive heart failure, uncontrolled diabetes mellitus, significant respiratory disease, or known immunosuppression;
* neurogenic bladder and/or sphincter abnormalities due to Parkinson's disease, multiple sclerosis, cerebral vascular accident, diabetes, etc.;
* a post void residual (PVR) volume above 250 ml measured by ultrasound or acute urinary retention
* compromised renal function (i.e., serum creatinine level above 1.8 mg/dl, or upper tract disease);
* confirmed or suspected bladder cancer;
* recent (within 3 months) cystolithiasis or hematuria;
* urethral strictures, bladder neck contracture, Urinary bladder stones
* or other potentially confounding bladder pathology;
* an active urinary tract infection.
* Enrolled in another treatment trial for any disease within the past 30 days.
* previous rectal surgery (other than hemorrhoidectomy) or history of rectal disease if the therapy may potentially cause injury to sites of previous rectal surgery, e.g., if a transrectal probe is used;
* previous pelvic irradiation or radical pelvic surgery;
* previous prostate surgery, balloon dilatation, stent implantation, laser prostatectomy, hyperthermia, or any other invasive treatment to the prostate
* Cancer that is not considered cured, except basal cell or squamous cell carcinoma of the skin (cured defined as no evidence of cancer within the past 5 years).
* Subject has an interest in future fertility and is not willing to undergo fertility treatments whatsoever.
* Any serious medical condition likely to impede successful completion of the study.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
IPSS | 6 months.
  Change of IPSS score by at least 3 points, in at least 75 % of the subjects, at 6 months follow-up.
  IPSS - The International Prostate Symptom Score. Scale: minimum 0 (zero), maximum 35. Lower values are better.
SAE | 5-7 days
  The incidence of unexpected serious adverse events related to Meditate iTind and/or implantation/retrieval procedures, as determined by the investigator and the study medical monitor.

SECONDARY OUTCOMES:
Urinary peak flow | 12 months
  Increase of maximal urinary peak flow

CONTACTS AND LOCATIONS:
Overall Officials: Claude Schulman, MD, Principal Investigator — Edith cavell clinic, Belgium
Locations (8):
- Belgium (2):
  - Edith Cavell, Brussels
  - Gent Hospital University, Ghent
- San Orbessano, Turin, Italy
- La Paz Hospital, Madrid, Spain
- Switzerland (2):
  - Kantonsspital Frauenfeld, Frauenfeld
  - Lausanne University Hospital, Lausanne
- United Kingdom (2):
  - Frimley Health NHS, London
  - University College Hospital, London

IPD SHARING:
Plan to Share IPD: No